CLINICAL TRIAL: NCT03207295
Title: A Randomized, Single-Blind, Placebo-Controlled, Single-Center Clinical Study of the Efficacy and Safety of Nesiritide on Early Postoperative Recovery After Total Cavo-Pulmonary Connection Surgery in Children
Brief Title: Impact of Nesiritide on Early Postoperative Recovery After Total Cavo-Pulmonary Connection Surgery in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Tibet Kang Zhe Pharmaceutical Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-898
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Congenital Heart Disease; Total Cavo-pulmonary Connection
Keywords: Nesiritide; Total Cavo-Pulmonary Connection; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Natriuretic Peptide, Brain; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention-Nesiritide (Experimental): A standard dose of Nesiritide(0.001ug/kg/min) is administered by a continuous infusion for ≥24 hours and ≤7 admission days after cardiac intensive care unit in postoperative children
  Interventions: Drug: Nesiritide
- Control-Normal saline (Placebo Comparator): Normal saline(2ml/h) is administered by a continuous infusion for ≥24 hours and ≤7 admission days after cardiac intensive care unit in postoperative children
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nesiritide — A standard dose of study drug was administered by a continuous infusion for ≥24 hours and ≤7 days after cardiac intensive care unit admission
  Arms: Intervention-Nesiritide
Drug: Normal saline — Normal saline(2ml/h) is administered by a continuous infusion for ≥24 hours and ≤7 admission days after cardiac intensive care unit in postoperative children
  Arms: Control-Normal saline

SUMMARY:
Nesiritide, a recombinant human B-type natriuretic peptide, has favorable effects on patient symptoms, hemodynamics, and the neurohumoral profile in adults with decompensated congestive heart failure and in those recovering from cardiac surgery involving cardiopulmonary bypass. Investigators seek to determine whether nesiritide would improve the early postoperative course after total cavo-pulmonary connection surgery in children.

DETAILED DESCRIPTION:
Objective: This study aims to evaluate the efficacy and safety of nesiritide after total cavo-pulmonary connection surgery in children. Investigators hypothesized that compared with placebo, patients assigned to receive nesiritide will improve early postoperative outcomes. Study design: The study is a a single-center, randomized, single-blinded, placebo-controlled, two-arm parallel-group clinical trial, patients undergoing total cavo-pulmonary connection surgery are assigned to receive nesiritide or placebo. A standard dose of study drug was administered by a continuous infusion for ≥24 hours and ≤7 days after cardiac intensive care unit admission. The primary outcome is days of chest drainage. Secondary outcomes included days of hospitalization measures of cardiovascular function, renal function, and adverse events and neurohumoral. The eligible participants will be allocated into intervention and control groups in a 1:1 ratio randomly. The intervention group will receive study drug. All the participants will be followed up during hospitalization .

Statistical analysis: Evaluation will be carried out on an intention-to-treat basis. Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. Elective general anesthesia down Fontan surgery patients, postoperative retention of patients with thoracic drainage tube
2. Age ≤ 14 years old between hospitalized patients, men and women are not limited
3. Postoperative hospital stay> 7 days
4. Patients or guardians voluntarily signed informed consent

Exclusion Criteria:

1. Before the group had serious head trauma need hospitalization or brain surgery patients
2. Who received organ transplants
3. Preoperative 48 hours application of recombinant B-type natriuretic peptide drugs
4. Preoperative cardiogenic shock or hypotension difficult to correct the patient
5. Preoperative patients with active arrhythmia
6. Preoperative serum creatinine> 1.5mg / dl or need dialysis patients
7. Preoperative liver dysfunction (glutamic oxalacetic transaminase /glutamic pyruvate transaminase elevated normal high 3 times or more)
8. Failed Fontan patients requiring secondary surgery
9. Patients with allergic to Nesiritide
10. The researchers believe that should not participate in the entry of patients
11. 3 months before the trial participated in other clinical trials

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Days of chest drainage | Up to 18 weeks
  Investigators will measure the daily chest drainage flow before discharge

SECONDARY OUTCOMES:
Days of hospitalization after surgery | Up to 20 weeks
  Postoperative hospital days
Postoperative early survival | The 30th day after surgery
  Number of days alive within 30 days of surgery.
Measures of heart rate | Baseline; Up to 20 weeks
  Investigators will measure the heart rate twice a day(Unit :beats per minute)
Measures of heart rhythm | Baseline; Up to 20 weeks
  Investigators will measure the heart rhythm twice a day
Measures of blood pressure | Baseline; Up to 20 weeks
  Investigators will measure the blood pressure twice a day(Units :mmHg)
Measures of central venous pressure | Up to 20 weeks
  Investigators will measure the central venous pressure(Unit :cmH2O)
Measures of liquid volume | Up to 20 weeks
  Investigators will measure the liquid volume each day after surgery
Measures of creatinine | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide;
  Investigators will measure the creatinine(Unit :umol/L)
Measures of blood urea nitrogen | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide;
  Investigators will measure the blood urea nitrogen(Unit :mmol/L)
Measures of glutamic oxalacetic transaminase | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide
  Investigators will measure the glutamic oxalacetic transaminase(Unit :U/L)
Measures of glutamic pyruvate transaminase | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide
  Investigators will measure the glutamic pyruvate transaminase(Unit :U/L)
Measures of total bilirubin | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide
  Investigators will measure the total bilirubin(Unit :umol/L)
Measures of N-terminal pro B-type natriuretic peptide | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide
  Investigators will measure the N-terminal pro B-type natriuretic peptide(Unit :pg/ml)
Measures of endothelin | Baseline; 1 day before using nesiritide; day 1 day 3 day 5 day 7 after using nesiritide
  Investigators will measure the endothelin(Unit :ng/L)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yajuan, MD,PhD, Principal Investigator — China National Center for Cardiovascular Disease; Duan Yabing, MD, Principal Investigator — China National Center for Cardiovascular Disease
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Consent for sharing of non identifiable study data for regulatory authorities